CLINICAL TRIAL: NCT03197701
Title: Maximal Effort-dependent Respiratory Flow Rates: Reproducibility and Reference Values
Brief Title: Maximal Effort-dependent Respiratory Flow Rates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 143201525127
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2016-09

CONDITIONS: Lung Function
Keywords: Lung function; Inspiratory flow rates

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The general objective of this project is to determine the best method to measure maximal inspiratory flow rates, to study their reproducibility and create reference equations in healthy subjects.

DETAILED DESCRIPTION:
1. Reproducibility and reference values in normal subjects: the investigators will propose a method for measurement of the maximal inspiratory flow rates (MIFR) and establish their reproducibility in normal subjects. The variability of these inspiratory flow rates will be compared with the variability of effort dependent and non-effort dependent expiratory flow rates.

   Also, reference equations will be drawn up and compared to the only existing set of reference values (2) (needing a revision).
2. Reproducibility in disease: the investigators will evaluate the reproducibility of the MIFR in patients with neuromuscular diseases (Steinert muscular dystrophy, amyotrophic lateral sclerosis) and with upper airway obstruction (tracheal stenosis, thyroid enlargement) and compare to the reproducibility of expiratory flow rates in this population.
3. Monitoring of diseases: In the neuromuscular patients MIFR will be correlated to the existing parameters used for monitoring of these diseases (respiratory muscle strength, forced vital capacity), with a longitudinal follow-up.

In the patients with upper airway obstruction the MIFR (quantitative measurement) will be compared to the visual inspection (qualitative interpretation) of the maximal flow-volume loop and also the evolution after a therapeutic intervention (airway stenting, thyroidectomy) will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* healthy hospital workers or visitors

Exclusion Criteria:

* current smokers or ex-smokers with a history of > 80 PY
* Presence or history of serious illness or thorax deformity (questionnaire)
* recent respiratory tract infection (1 week)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Normal values for maximal inspiratory flow rates | 3 years
  Peak inspiratory flow rate (PIF)
Normal values for maximal inspiratory flow rates | 3 years
  Maximal flow rate when 50% of inspiratory vital capacity has been inhaled (FIF50)

SECONDARY OUTCOMES:
Reproducibility of maximal inspiratory flow rates | 3 years
  Coefficient of variation for peak inspiratory flow rate (PIF)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Hanon, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No